CLINICAL TRIAL: NCT04103593
Title: Effects of 12-weeks of High-intensity Resistance Aerobic Circuit Exercise Training on Epigenetic Aging and Inflammation in Older HIV-infected Veterans
Brief Title: Functional Interval Training for Veterans Exercising Through Telehealth.
Acronym: FIT-VET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Atlanta VA Medical Center (U.S. Federal Agency); Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: F2790-R
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: HIV Infection
Keywords: exercise training; video telehealth; DNA methylation; Aging; HIV
MeSH Terms: conditions — HIV Infections | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise trial of 12-weeks high-intensity circuit exercise delivered by VTEL to older Veterans living with HIV that compares exercise group to standard of care sedentary control group
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise group (Experimental): High-intensity circuit exercise training will be performed 3 times weekly for 12 weeks in a group setting. Circuit training is an exercise modality consisting of a series of exercises at different stations. Exercise training will be delivered by VTEL broadcast from the Salem VAMC to participants at the Atlanta VAMC and Baltimore VAMC. Rooms will be equipped with steps, hand and ankle weights, dumbbells, chairs and bands. No stationary exercise equipment will be used in either AEX or RT.
  Interventions: Behavioral: exercise training
- control group (No Intervention): Sedentary activity (confirmed at eligibility no more than 1 structured physical activity/week) will be continued in participants randomized to the control group. Participants have the option after 12-week intervention phase to enter "delayed" exercise training to assure that all participants can receive exercise training.

INTERVENTIONS:
Behavioral: exercise training — 12-weeks of high-intensity functional circuit exercise that will be broadcasted from the Salem VAMC to older Veterans living with HIV in the Atlanta and Baltimore VAMCs
  Arms: exercise group

SUMMARY:
Most Veterans living with HIV are 50 years of age or older and can expect to live more than 20 years longer with HIV medication. However, despite this success, Veterans living with HIV are more likely to have age-related diseases and loss of fitness and muscle that place them at increased risk for disability. This is a major priority for the VHA, the largest provider of HIV care in the United States. The goal of this study is to test a circuit exercise program in Veterans living with HIV that is designed to slowdown the aging process. The exercise program will be widely available by Video Teleconferencing (VTEL) and does not require stationary exercise equipment, making it widely accessible. This research will help reach the goal for Veterans to preserve their quality of life and ability to function independently. Novel findings will strengthen strategies to maintain life-long fitness through a personalized exercise prescription.

DETAILED DESCRIPTION:
The Veterans Health Administration (VHA) is the largest U.S. HIV health provider with 64% of these Veterans 50+ years of age. HIV infection in the setting of antiretroviral therapy represents a chronic disease with an advanced aging phenotype manifested as increased cardiovascular disease, sarcopenia, and frailty, primarily driven by systemic inflammation. The investigators found a 42% reduction in VO2peak in older HIV+ adults that significantly improved with high-intensity aerobic (AEX) and resistance training (RT). Yet, durable strategies for high-intensity exercise in older adults remain a challenge and limited data are available in older HIV+ adults. There is an urgent need to address these knowledge gaps in order to prevent widespread disability in HIV+ Veterans. The objective is to provide a high-intensity exercise program for older Veterans that can be widely disseminated and attenuates processes underlying aging. Epigenetic changes with increased age encapsulate the putative effects of biological aging and lifestyle factors. DNA methylation (DNAm) patterns are frequently modified in genes encoding pro-inflammatory cytokines, but can be reversed with exercise training. DNA methylation age (DNAm Age) is an epigenetic biomarker that is expressed in years and provides a concrete benchmark of advanced aging. The investigators found that HIV+ adults have DNAm Age 11 years greater than age-matched adults without HIV. Further, in adults without HIV, increased DNAm Age is associated with physical inactivity, weakness and frailty. Preliminary data in the Veterans Aging Cohort Study (VACS) show that DNAm Age correlates with the VACS Index, a measure of frailty in HIV+ adults. However, the impact of exercise training on DNAm Age has yet to be determined in any patient population. The investigators propose to adapt center-based high-intensity AEX+RT intervention in older HIV+ Veterans into a video telehealth (VTEL) delivered functional (no stationary equipment) exercise program that leverages epigenetic outcomes to demonstrate anti-aging effects of exercise. The overarching hypothesis is that VTEL high-intensity functional circuit exercise in older HIV+ Veterans will improve the advanced aging phenotype and attenuate DNAm epigenetic processes underlying aging. Experimental approach includes a 12-week VTEL exercise intervention in 80 older HIV+ Veterans who are randomized to exercise or standard of care sedentary control groups. AIM 1 will determine the effect of VTEL exercise on VO2peak, sarcopenia, and frailty as phenotypic outcomes of advanced aging in HIV. AIM 2 will investigate the effect of VTEL exercise on DNAm Age as a biomarker of advanced aging. AIM 3 will determine the effect of VTEL exercise on DNA methylation of specific genes encoding specific pro-inflammatory cytokines in leukocytes. This approach will advance an understanding of effective and feasible exercise strategies to prevent and minimize disability in patient populations with advanced aging. Findings will provide an innovative approach to functional exercise in all older adults. DNAm Age could be used as a personalized benchmark for an individual's benefit from exercise to promote sustainable behavior change. Findings will also provide epigenetic risk profiles that can be used to generate a personalized exercise prescription, an important next step in the next decade of precision medicine. The proposal leverages exercise training experience in HIV and VTEL, availability of 3,000 HIV+ Veterans at Atlanta and Baltimore VAMCs, and the VHA VTEL infrastructure. The capacity to disseminate VTEL exercise with minimal cost using existing infrastructure will facilitate large-scale dissemination and national impact. Deliverables include improved clinical outcomes and substantial cost savings from reduced hospitalization and institutionalization rates.

ELIGIBILITY:
Inclusion Criteria:

* Veteran living with HIV and under care at VAMC
* 50 years of age and older
* Stable antiretroviral therapy (same ARV medications within 3 months)
* At least one HIV-1 PCR < 20 c/ml (viral load) within prior 6 months

Exclusion Criteria:

* History of AIDS defining illnesses (within 6 months; CDC Criteria)
* Myocardial infarction (within 3 months)
* Exertional or unstable angina (current chest pain that limits activity)
* Severe congestive heart failure (EF < 20% in last year or NYHA Classification III or IV)
* Uncontrolled hypertension (SBP >180 &/or DBP > 110 mm Hg)
* Therapy with beta blockers or non-dihydropyridine calcium channel blocker (within 1 month)
* Screening EKG with ischemia, complex arrhythmia, or high-grade block (per Minnesota Code)
* Poorly controlled DM within prior 1 month (FBS>180 mg/dl, RBS > 299 mg/dl, or HbA1C > 10)
* Receiving treatment for cancer except skin cancer (within 3 months)
* Peripheral vascular disease with claudication
* Severe arthritis limiting ambulation
* Neurologic disease limiting ambulation (requiring assist device)
* End stage liver disease (decompensated liver disease)
* Chronic renal failure (requiring dialysis)
* Severe pulmonary disease (home O2, admission for dyspnea or pneumonia within 1 month)
* Use of systemic steroids (testosterone or glucocorticoids) or growth hormone (within 6 months)
* Dementia (based on Evaluation to Consent)
* Signs or symptoms of any medical comorbidity that would preclude exercise testing or training
* Exercise on routine basis (structured aerobic exercise > 3 times per week) within 1 month
* Past medical history of COPD or emphysema AND mMRC score =4

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris Ann K Oursler, MD, Principal Investigator — Salem VA Medical Center, Salem, VA; Vincent Marconi, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA; Alice S. Ryan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (3):
- United States (3):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Salem VA Medical Center, Salem, VA, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.

REFERENCES:
- [Background] Oursler KK, Marconi VC, Wang Z, Xu K, Montano M, So-Armah K, Justice AC, Sun YV. Epigenetic Age Acceleration Markers Are Associated With Physiologic Frailty and All-Cause Mortality in People With Human Immunodeficiency Virus. Clin Infect Dis. 2023 Feb 8;76(3):e638-e644. doi: 10.1093/cid/ciac656. PMID 35970820
- [Background] Oursler KK, Marconi VC, Briggs BC, Sorkin JD, Ryan AS; FIT VET Project Team. Telehealth Exercise Intervention in Older Adults With HIV: Protocol of a Multisite Randomized Trial. J Assoc Nurses AIDS Care. 2022 Mar-Apr 01;33(2):168-177. doi: 10.1097/JNC.0000000000000235. PMID 33481463
- [Result] Oursler KK, Briggs BC, Lozano AJ, Harris NM, Parashar A, Ryan AS, Marconi VC; for the FIT VET Project Team. Association of chronotropic incompetence with reduced cardiorespiratory fitness in older adults with HIV. AIDS. 2024 May 1;38(6):825-833. doi: 10.1097/QAD.0000000000003840. Epub 2024 Jan 11. PMID 38578959
- [Result] Oursler KK, Briggs BC, Lozano AJ, Harris NM, Marconi VC, Ryan AS. Association of Step Count with Cardiorespiratory Fitness: Results from the Virtual 2-Minute Step Test. Arch Rehabil Res Clin Transl. 2024 Dec 9;6(4):100369. doi: 10.1016/j.arrct.2024.100369. eCollection 2024 Dec. PMID 39822200

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Group | Control Group
Started | 45 | 44
Completed | 31 | 36
Not Completed | 14 | 8

BASELINE CHARACTERISTICS:
Population: Participants randomized into the exercise and control arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Control Group | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 27 | 57
  >=65 years | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (6.6) | 63.1 (7.5) | 62.9 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 43 | 43 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 44 | 44 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 39 | 78
  White | 5 | 4 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 44 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline VO2peak to After 12-week Exercise Intervention
Description: O2 consumption at peak exercise effort, VO2peak, is used as the standard measure of aerobic capacity in sedentary adults since the majority are not able to reach maximal aerobic capacity defined as a plateau in O2 consumption. VO2peak will be the average of the final 30 second values of O2 consumption at peak exercise on a treadmill using a modified Bruce protocol
Time Frame: baseline and 13-weeks
Population: Only participants who completed 12-week follow up testing. Among completers, 2 were missing VO2 data at Follow Up; Baseline data was provided for these participants.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 31 | 36
Liters/minute
  Baseline | 1.99 (0.46) | 2.05 (0.57)
  12 Week Follow Up: number analyzed (Participants) | 30 | 35
  12 Week Follow Up | 2.07 (0.53) | 2.07 (0.47)
  Change: number analyzed (Participants) | 30 | 35
  Change | 0.09 (0.23) | 0.00 (0.29)

2. Secondary Outcome: Change From Baseline DNA Methylation to After 12-week Exercise Intervention
Description: Epigenome-wide association studies (EWAS)
Time Frame: baseline and 13-weeks
Reporting Status: Not Posted, anticipated posting 2026-06

3. Other Pre Specified Outcome: VTEL Exercise Training Feasibility
Description: Rates will be calculated for enrollment, attendance, and retention
Time Frame: through study completion, an average of 1 year
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: From consent to follow up testing (up to 1.5 years or as needed)
Description: Not different
Arm/Group | Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 1/44
Serious Adverse Events (participants affected / at risk) | 1/45 | 2/44
Other Adverse Events (participants affected / at risk) | 28/45 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise Group (N=45) | Control Group (N=44)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalization for large bowel perforation
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hospitalization for community-acquired pneumonia
Hospitalization (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hospitalization for hyperthyroidism
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise Group (N=45) | Control Group (N=44)
COVID exposure (Infections and infestations) | 1 (1) | 0 (0)
Injury from a fall (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Cardiac disorders) | 2 (2) | 0 (0)
Hip and leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Hypertensive episode (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arm weakness (Nervous system disorders) | 1 (1) | 0 (0) — Existing cervical spine problem
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Irregular heart rate (Cardiac disorders) | 4 (4) | 0 (0) — Tachycardia, high HR
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Oral surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Upset stomach/vomiting/diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Wrist pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Injury from car crash (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness/low blood sugar related to diabetes (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee pain from arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0) — Chest pain or tightness during exercise
Cold/flu symptoms (Infections and infestations) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT04103593/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT04103593/ICF_002.pdf